CLINICAL TRIAL: NCT00300404
Title: Effect of Add-on Anti-Toxoplasmosis Treatment on Parameters Defining Toxoplasma Gondii Infection and on Psychopathology in Patients With Schizophrenia or Major Depression Serologically Positive for Toxoplasma Gondii - Phase 3 Study
Brief Title: Effect of Specific Anti-Toxoplasmatic Add-on Medication in Toxoplasma Gondii Seropositive Individuals With Schizophrenia or Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zentrum für Integrative Psychiatrie (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOXO-KI-TT; SMRI grant # 01T-404
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2006-05-22 (Estimated); Status verified 2006-03

CONDITIONS: Schizophrenia; Major Depression
Keywords: Schizophrenia; Psychosis; Depression; Affective Disorder
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Psychotic Disorders; Depression; Mood Disorders | interventions — Pyrimethamine; Leucovorin

INTERVENTIONS:
Drug: daraprim
Drug: pyrimethamine
Drug: folinic acid

SUMMARY:
We investigate whether the add-on specific antitoxoplasmatic medication has positive effects in individuals with schizophrenia or major depression seropositive for Toxoplasma gondii (TG) infection. As TG modulates neurotransmitter metabolism affecting serotonin and dopamine we hypothesize that this chronic persistent infection might play a role for depressive and psychotic symptomatology. Therefore, on the basis of an ex juvantibus approach, specific anti TG medication might further improve psychiatric symptomatology in affected patients. This is investigated in a double-blind, placebo-controlled, randomized treatment trial.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or Major Depression
* Both genders
* Adult
* Patients are able to give informed consent

Exclusion Criteria:

* Additional diagnosis of substance abuse/dependency
* Continuous treatment with medication not compatible with study medication
* Medical status not compatible with study medication
* Any condition that increases study risk considerably
* Pregnancy, nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-01; Study Completion 2005-09

PRIMARY OUTCOMES:
Psychopathology ratings

SECONDARY OUTCOMES:
TG infection parameters

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Hinze-Selch, MD, Principal Investigator — Zentrum für Integrative Psychiatrie